CLINICAL TRIAL: NCT00045799
Title: Safety & Efficacy of Omeprazole Sodium Bicarbonate for the Prevention of Upper GI Bleeding in the Critically Ill
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OSB-IR C03
Record Dates: First submitted 2002-09-09; First posted 2002-09-11 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole sodium bicarbonate immediate release PWD/FS (Experimental)
  Interventions: Drug: Omeprazole sodium bicarbonate immediate release PWD/FS
- Cimetidine IV (Active Comparator)
  Interventions: Drug: Cimetidine IV

INTERVENTIONS:
Drug: Omeprazole sodium bicarbonate immediate release PWD/FS
  Arms: Omeprazole sodium bicarbonate immediate release PWD/FS
Drug: Cimetidine IV
  Arms: Cimetidine IV

SUMMARY:
Critically ill patients are at an increased risk of having upper gastrointestinal (GI) bleeding due to stress related mucosal damage. Cimetidine, delivered continuously through intravenous infusion, is the only drug that the FDA has approved for the prevention of upper GI bleeding in critically ill patients. The present trial is intended to assess the safety and efficacy of an omeprazole sodium bicarbonate immediate-release suspension in this indication.

DETAILED DESCRIPTION:
This trial will be a triple-blind, double-dummy, prospective, multicenter, randomized clinical trial comparing the effectiveness of OSB-IR to the effectiveness of intravenous cimetidine in preventing upper GI bleeding at risk for SRMD.

ELIGIBILITY:
Patients will be included in the trial if they meet all of the following criteria:

1. An adult or adolescent (greater than or equal to 16 years of age) male or non-pregnant female requiring mechanical ventilation for greater than or equal to 48 hours.
2. An anticipated ICU stay of greater than or equal to 72 hours.
3. An Acute Physiology and Chronic Health Evaluation (APACHE II) score of >11 immediately before randomization.
4. At least one other risk factor for upper GI bleeding due to stress-related mucosal damage in addition to mechanical ventilation. Acceptable "other" risk factors include:

   * closed-head injury
   * multiple trauma to head, chest, abdomen, solid organs, or limbs
   * major surgical procedures (eg, mastectomy, pancreatectomy, cardiovascular surgery) 24 hours previous to screening
   * extensive burns (greater than or equal to 30% of the body surface area)
   * acute renal failure (urine output <0.5 mL/kg of body weight/hr for one hour, despite adequate fluid resuscitation)
   * acid-base disorder (pH less than or equal to 7.3 or base deficit greater than or equal to 5.0 mMol/L with a plasma lactate level >1.5 times the upper limit of normal for the reporting laboratory)
   * coagulopathy (a platelet count <50,000/mm3, an INR of >1.5 [i.e., prothrombin time >1.5 times the control value], or a partial-thromboplastin time >2.0 times the control value)
   * marked jaundice (defined as plasma total bilirubin concentration of >51.3 micromol/L or >3 mg/dL)
   * coma
   * hypotension (either a systolic blood pressure <80 mm Hg for 2 hours or more or a decrease of greater than or equal to 30 mm Hg in the systolic blood pressure)
   * shock (arterial blood pressure less than or equal to 90 mm Hg or mean arterial pressure less than or equal to 70 mm Hg for at least one hour despite adequate fluid resuscitation, adequate intravascular volume status or the use of vasopressors in an attempt to maintain a systolic blood pressure of greater than or equal to 90 mm Hg or a mean arterial pressure of greater than or equal to 70 mm Hg)
   * sepsis (defined as a positively cultured or clinically diagnosed infection with at least three of the following: a body temperature of greater than or equal to 38 degrees C [greater than or equal to 100.4 degrees F] or less than or equal to 36 degrees C [less than or equal to 96.8 degrees F], a heart rate of greater than or equal to 90 beats/min, tachypnea manifested by a respiratory rate of greater than or equal to 20 breaths/min, or hyperventilation as indicated by a PaCO2 of less than or equal to 32 mm Hg, and a white blood cell count of greater than or equal to 12,000 cells/mm3 or less than or equal to 4,000 cells/mm3, or the presence of >10% bands)
5. An intact stomach and a nasogastric or an orogastric tube in place.
6. An anticipation of no enteral feedings for the first two days of trial drug treatment.

Exclusion Criteria

Patients will be excluded from trial participation if they meet any of the following criteria:

1. A status of "No Cardiopulmonary Resuscitation (CPR)".
2. If >48 hours has elapsed since the patient became eligible for the trial.
3. Known history of vagotomy, pyloroplasty, gastroplasty, or any other gastric surgery.
4. Known allergy to cimetidine or omeprazole.
5. Active GI bleeding (including esophageal and gastric variceal bleeding, duodenal and gastric ulcers).
6. Significant risk of swallowing blood (i.e., severe facial trauma, oral lacerations, hemoptysis).
7. Enteral feedings for the first two days of trial drug treatment.
8. Use of an investigational drug within 30 days prior to randomization.
9. Critical/intensive care unit admission following esophageal, gastric, or duodenal surgery or trauma.
10. Known history of upper gastrointestinal lesions that are likely to bleed (e.g., esophageal or gastric varices, gastric polyps, tumors, etc. but excluding patients with gastric or duodenal ulcer disease).
11. Any medical or surgical condition that precludes administration of an oral medication (i.e., OSB-IR).
12. End stage liver disease.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2002-05; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (58):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Maricopa Medical Center, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Ltd, Phoenix, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - Providence St. Joseph's Medical Center, Burbank, California
  - Verdugo Hills Hospital, Burbank, California
  - Loma Linda Medical Center, Loma Linda, California
  - Stanford University School of Medicine, Stanford, California
  - Christiana Hospital, Newark, Delaware
  - PAB Clinical Research, Brandon, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Miami VAMC, Miami, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - USF Pulmonary Research, Tampa, Florida
  - Protocare Trials, Austell, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Protocare - Alexian Brothers Center for Clinical Research, Elk Grove Village, Illinois
  - West Suburban Hospital, Oak Park, Illinois
  - University of Iowa Health Care, Iowa City, Iowa
  - Department of Medicine, Kansas City, Kansas
  - Medical Center of LA at New Orleans (LSU Health Sci Ctr), New Orleans, Louisiana
  - Louisiana State University, Shreveport, Louisiana
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Truman Medical Center Hospital Hill, Kansas City, Missouri
  - St. Johns Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Cooper Hospital/UMC, Camden, New Jersey
  - Trinitas Hospital, Elizabeth, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - University Hospital, Newark, New Jersey
  - SUNY Health Science Center, Brooklyn, New York
  - Winthrop University Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - St. Vincent's Catholic Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Akron General Hospital, Akron, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - North Texas Affiliated Medical Group, Fort Worth, Texas
  - Texas Tech University Health Sciences Center, Odessa, Texas
  - University of Vermont, Burlington, Vermont
  - Pulmonary & Critical Care, Richmond, Virginia
  - West Virginia University Hospitals, Inc, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin